CLINICAL TRIAL: NCT04760548
Title: Segmentation of Structural Abnormalities in Chronic Lung Diseases
Acronym: NOVAA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hôpital Haut Lévêque (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Collaborative NOVAA study group (Unknown)
Responsible Party: Sponsor-Investigator, Hôpital Haut Lévêque, Director, Hôpital Haut-Lévêque
Organization: Hôpital Haut-Lévêque (Other)
Other Study IDs: NOVAA
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-09

CONDITIONS: Cystic Fibrosis; Asthma; COPD; Interstitial Lung Disease
MeSH Terms: conditions — Cystic Fibrosis; Asthma; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Train dataset: This group is dedicated to developing an automated algorithm
  Interventions: Other: Observational study
- Test dataset: This group is dedicated to testing the semantic performance of an automated algorithm
  Interventions: Other: Observational study
- Clinical Validations: Patients groups are dedicated to assessing the clinical validity of the measurement in independent validation cohorts, with or without longitudinal evaluations such as monitoring of a treatment effect
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study

SUMMARY:
Lung structural abnormalities are complex, time-consuming, and may lack reproducibility to evaluate visually on CT scans. The study's aim is to perform automated recognition of structural abnormalities in CT scans of patients with chronic lung diseases by using dedicated software.

DETAILED DESCRIPTION:
Three chronic lung diseases will constitute the target of the study, by using retrospective data from each lung disease:

* Cystic fibrosis
* Asthma and COPD
* Interstitial lung diseases

Dedicated algorithms will be developped for each disease condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic lung disease and clinical examination, pulmonary function test, and CT acquired during a routine follow-up

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic lung disease and a Clinical examination, pulmonary function test, and CT acquired during an annual routine follow-up
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2024-02-17 (Estimated); Study Completion 2024-02-17 (Estimated)

PRIMARY OUTCOMES:
Validity of automated measurement | From date of inclusion until the date of final quantification, assessed up to 12 months
  Correlations and comparisons with other biomarker of the disease severity

SECONDARY OUTCOMES:
Correlation with pulmonary function test | From date of inclusion until the date of final quantification, assessed up to 12 months
  Correlation of quantitative measurement with pulmonary function
Longitudinal variation over time | From date of inclusion until the date of final quantification, assessed up to 12 months
  Comparison of quantitative measurement at two time points
Reproducibility | From date of inclusion until the date of final quantification, assessed up to 12 months
  Evaluation of measurements when performed twice

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Berger, Pr, Study Chair — Hopital Haut Leveque
Locations (1):
- Hopital Haut Leveque, Pessac, France

IPD SHARING:
Plan to Share IPD: Undecided
Automated software measurements

REFERENCES:
- [Derived] Dournes G, Hall CS, Willmering MM, Brody AS, Macey J, Bui S, Denis de Senneville B, Berger P, Laurent F, Benlala I, Woods JC. Artificial intelligence in computed tomography for quantifying lung changes in the era of CFTR modulators. Eur Respir J. 2022 Mar 3;59(3):2100844. doi: 10.1183/13993003.00844-2021. Print 2022 Mar. PMID 34266943